CLINICAL TRIAL: NCT02210481
Title: Impact of Intravitreal Glucose Rate in Macular Thinning Following Retinal Detachment or Epimacular Membrane Surgery
Brief Title: The Role of Intravitreal Glucose in Macular Thinning Following Surgery for Retinal Detachment or Epimacular Membrane
Acronym: GLU-MAC
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: AOL2010-02
Record Dates: First submitted 2014-08-05; First posted 2014-08-06 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Vitrectomy; Macular Thinning
Keywords: vitrectomy,; macular thinning,; retinal detachment,; epimacular membrane,; intravitreal glucose,; OCT
MeSH Terms: conditions — Retinal Detachment; Epiretinal Membrane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GLUC-MAC-COHORT: post vitrectomy for retinal detachment or epimacular membrane patients

SUMMARY:
Comparison between intravitreous glucose rate and macular thinning measured by Ocular Coherence Tomography (OCT) at 3 months post vitrectomy for retinal detachment or epimacular membrane. Hypothesis : Association between post-operative macular thickness and intravitreous glucose rate

DETAILED DESCRIPTION:
Comparison between intravitreous glucose rate and macular thinning measured by OCT at 3 months post vitrectomy for retinal detachment or epimacular membrane. The cohort is divided in 2 groups, one with the thinnest macular measurement under 190µm, and the others above 190µm. We are looking for a correlation between increasing glucose rates and decreased macular thickness.

ELIGIBILITY:
Inclusion Criteria:

* patient who underwent vitrectomy for retinal detachment or epimacular membrane

Exclusion Criteria:

* patient suffering of diabetes,
* recurrence of retinal detachment,
* age-related macular degeneration,
* post surgical macular oedema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cohort composed of patients undergoing vitrectomy for retinal detachment or epimacular membrane at Reims University Hospital
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
macular thickness measured by OCT | 3 months post-operatively

SECONDARY OUTCOMES:
visual acuity | 3 months post-operatively

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Reims, Reims, France